CLINICAL TRIAL: NCT02001337
Title: Examination of the Pancreas in New-onset Diabetes (EXPAND Study)
Brief Title: Examination of the Pancreas in New-onset Diabetes
Acronym: EXPAND
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gloria M. Petersen, Principal Investigator, Mayo Clinic
Other Study IDs: 10-006868
Record Dates: First submitted 2013-11-22; First posted 2013-12-04 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus
Keywords: pancreatic cancer; new-onset diabetic; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Pancreatic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 60ml of whole blood. 5ml urine sample for pregancy testing (if necessary). Stool and saliva samples may be collected.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: medical chart review — baseline, quarterly follow-up for 24 months
Other: survey administration — baseline
Other: Specimen collection — baseline

SUMMARY:
The purpose of this study is to create a prospective cohort of subjects with increased probability of being diagnosed with pancreatic cancer and then screen this cohort for pancreatic cancer

DETAILED DESCRIPTION:
Compared to the general population, subjects >50 years of age with new-onset diabetes (DM) are 8-times more likely to have pancreatic cancer (PaC). The likelihood of PaC in new-onset DM is further increased in those who have weight loss or elevated CA19-9. In this study patients with newly diagnosed diabetes will be prospectively identified. Those with weight loss and/or elevated pancreatic cancer marker (CA 19-9) will undergo pancreatic imaging. All subjects will be followed up to 24 months. If successful in identifying surgically removable PaC, this study will fundamentally change our practice and will be a major breakthrough in PaC treatment and research.

ELIGIBILITY:
Patient Characteristics:

--Suspected or definite new-onset diabetes based on recent blood sugar and hemoglobin A1c values

* No acute illness or steroid therapy
* No prior pancreas surgery

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected or definite new-onset diabetes
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2013-05; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
To create a prospective cohort of subjects with increased probability of being diagnosed with pancreatic cancer and identify pancreatic cancer in this cohort. | Follow subjects for 2 years.
  We will prospectively identify patients with newly diagnosed diabetes and perform pancreatic imaging to identify pancreatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Petersen, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials